CLINICAL TRIAL: NCT00655018
Title: Lifestyle Intervention and Antioxidants in Children With Nonalcoholic Fatty Liver Disease: A Randomized, Controlled Trial
Brief Title: Effect of Vitamin E on Pediatric Nonalcoholic Fatty Liver Disease (NAFLD)
Acronym: VITENAFLD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Valerio Nobili, MD, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITENAFLD
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-03

CONDITIONS: Inflammation; Fibrosis; Insulin Resistance
Keywords: Non-Alcoholic Fatty Liver Disease (NAFLD); Non-Alcoholic Steatohepatitis (NASH); Liver histology; Insulin Resistance; Weight loss; Alpha-tocopherol; ascorbic acid
MeSH Terms: conditions — Inflammation; Fibrosis; Insulin Resistance; Non-alcoholic Fatty Liver Disease; Weight Loss | interventions — alpha-Tocopherol; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin group (Experimental): alpha tocopherol 600 IU/d plus ascorbic acid 500 mg/d and lifestyle intervention [hypocaloric Diet(25-30 cal/kg/d) or isocaloric (40-45 cal/kg/d) and physical activity].
  Interventions: Dietary Supplement: Vitamin treatment (alpha tocopherol plus ascorbic acid)
- 2 (Placebo Comparator): placebo and lifestyle intervention [hypocaloric Diet(25-30 cal/kg/d) or isocaloric (40-45 cal/kg/d) and physical activity].
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin treatment (alpha tocopherol plus ascorbic acid) — alpha tocopherol 600 IU/d plus ascorbic acid 500 mg/d and lifestyle intervention [hypocaloric Diet(25-30 cal/kg/d) or isocaloric (40-45 cal/kg/d) and physical activity].
  Other Names: alpha-tocoferol
  Arms: Vitamin group
Dietary Supplement: Placebo — placebo and lifestyle intervention [hypocaloric Diet(25-30 cal/kg/d) or isocaloric (40-45 cal/kg/d) and physical activity].
  Arms: 2

SUMMARY:
No proven treatment exists for nonalcoholic fatty liver disease (NAFLD) in children and adolescents. We aim to determine the efficacy of lifestyle intervention with or without antioxidant therapy in pediatric NAFLD.

DETAILED DESCRIPTION:
InChildren or adolescents with well-characterized and liver biopsy confirmed NAFLD will be enrolled. They will be randomized to treatment with alpha tocopherol 600 IU/d plus ascorbic acid 500 mg/d (n=45) or an identical placebo (n=45) given orally. All patients will be included in a lifestyle intervention program consisting of a diet tailored on the individual requirements and physical exercise. The body mass index (BMI) and BMI Z-score will be calculated . Obesity was defined for a percentile of BMI ≥ 95th percentile for age and gender .

Patients will undergo a medical evaluation every three months during the 24-month study period. Laboratory tests including liver enzymes and lipids will be repeated at 3-month intervals during the 24-month study duration. Ultrasonography of the liver will be repeated at the end of the study period.

Evaluation of Glucose Metabolism and Insulin Sensitivity A 2-hour oral glucose tolerance test (OGTT) will be performed at baseline and repeated at 24 mo. of treatment with the standard 1.75 g of glucose per kg, or maximum of 75 g. Glucose tolerance status will be determined according to the classification of the American Diabetes Association in which fasting plasma glucose (FPG) levels up to 99 mg/dl are considered normal; impaired fasting glucose (IFG) is defined by a FPG of 100-125 mg/dl; impaired glucose tolerance (IGT) is defined by a 2-hour plasma glucose of 140-199 mg/dl; diabetes mellitus is defined by a FPG ≥126 mg/dl, or a 2-hour plasma glucose ≥200 mg/dl .

The degrees of insulin resistance and sensitivity will be determined, respectively, by the homeostatic model assessment (HOMA-IR) using the formula: IR = (insulin*glucose)/22.5; and by the insulin sensitivity index (ISI) derived from OGTT using the formula: ISI = (10,000/square root of [fasting glucose x fasting insulin] x [mean glucose x mean insulin during OGTT]).

Liver biopsy Liver biopsy will be performed at baseline and repeated at 24 mo. of treatment. Biopsies will be routinely processed and analyzed as described previously. Pre- and post-treatment liver biopsies will be reviewed and scored by a single pathologist who will be unaware of the assigned treatment, patients' clinical and laboratory data, and liver biopsy sequence. The main histological features of NAFLD including steatosis (macro and microvesicular), inflammation (portal and lobular), hepatocyte ballooning, and fibrosis will be scored using the scoring system for NAFLD recently proposed by the NIH-sponsored NASH Clinical Research Network.

ELIGIBILITY:
Inclusion Criteria:

* persistently elevated serum aminotransferase levels,
* diffusely echogenic liver on imaging studies suggestive of fatty liver, and
* biopsy consistent with the diagnosis of NAFLD.

Exclusion Criteria:

* hepatic virus infections (HCV RNA-PCR negative),
* Hepatitis A, B, C, D, E and G,
* cytomegalovirus and Epstein-Barr virus,
* alcohol consumption,
* history of parenteral nutrition,
* and use of drugs known to induce steatosis (e.g. valproate, amiodarone or prednisone) or to affect body weight and carbohydrate metabolism.
* Autoimmune liver disease, metabolic liver disease, Wilson's disease, and a-1-antitrypsin-associated liver disease were ruled out using standard clinical, laboratory and histological criteria.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2003-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
serum levels of aminotransferases | months 12 and 24

SECONDARY OUTCOMES:
Liver histology (inflammation and fibrosis) | month 24

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Nobili, MD, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (1):
- Dept. Of HepatoGastoEnterology and Nutrition, Liver Unit, Rome, Italy

REFERENCES:
- [Background] Bugianesi E, Gentilcore E, Manini R, Natale S, Vanni E, Villanova N, David E, Rizzetto M, Marchesini G. A randomized controlled trial of metformin versus vitamin E or prescriptive diet in nonalcoholic fatty liver disease. Am J Gastroenterol. 2005 May;100(5):1082-90. doi: 10.1111/j.1572-0241.2005.41583.x. PMID 15842582
- [Background] Vajro P, Mandato C, Franzese A, Ciccimarra E, Lucariello S, Savoia M, Capuano G, Migliaro F. Vitamin E treatment in pediatric obesity-related liver disease: a randomized study. J Pediatr Gastroenterol Nutr. 2004 Jan;38(1):48-55. doi: 10.1097/00005176-200401000-00012. PMID 14676594
- [Background] Lavine JE. Vitamin E treatment of nonalcoholic steatohepatitis in children: a pilot study. J Pediatr. 2000 Jun;136(6):734-8. PMID 10839868
- [Result] Nobili V, Manco M, Devito R, Ciampalini P, Piemonte F, Marcellini M. Effect of vitamin E on aminotransferase levels and insulin resistance in children with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2006 Dec;24(11-12):1553-61. doi: 10.1111/j.1365-2036.2006.03161.x. PMID 17206944
- See also: Hospital's web site — http://www.ospedalebambinogesu.it/